CLINICAL TRIAL: NCT03512925
Title: Effects of a Standardized Post-coercion Review Session on Objective and Perceived Coercion
Brief Title: Effects of a Standardized Post-coercion Review Session.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Federal Ministry of Health, Germany (Other Government)
Responsible Party: Principal Investigator, Alexandre Wullschleger, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NBZM_MZ
Record Dates: First submitted 2018-01-30; First posted 2018-05-01 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Coercive Measures
Keywords: Coercion; Post-coercion review; Mental health; Seclusion; Mechanical restraint
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Eligible participants are randomly assigned either to the intervention arm (standardized post-coercion review session session) or to the Treatment-as-usual (TAU) arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized post-coercion review (Experimental): Intervention: Standardized post-coercion review session. Patients allocated to this arm receive a standardized post-coercion review of the coercive measure they experienced using the developed guidelines.
  Interventions: Other: Standardized debriefing session of coercive measures
- Control group (No Intervention): Patients allocated to this arm are treated following usual standards and routine. This might include some form of post-coercion review that doesn't follow the developed standardized guidelines.

INTERVENTIONS:
Other: Standardized debriefing session of coercive measures — Debriefing session following the developed guidelines including setting and themes.
  Arms: Standardized post-coercion review

SUMMARY:
The present study aims at exploring the impact of a standardized post-coercion review session of coercive measures that took place in the psychiatric inpatient setting in reducing the use of coercive measures and the subjective perception of coercion. It is well known that coercive measures have a major negative impact on the health, well-being and the course of treatment of patients suffering from mental health issues. Many interventions have been implemented in the last years to reduce the use of coercion and limit its consequences.

The investigators developed a standardized post-coercion review intervention. This session takes place as soon as possible after the concerned coercive measure and is moderated by a member of staff who has not been involved in the use of coercion. Other persons involved are the patient, a staff member who took the decision leading to the use of the coercive measure, and a one of the patient's relatives.

Hypothesis is that the use of this standardized intervention can reduce the use of subsequent coercive measures and level of perceived coercion, prevent the development of post-traumatic symptoms, help preserving a trustful therapeutic relationship and positively change the attitude of staff regarding the use of coercion. This intervention has been proven to be well accepted by patients and staff members in a previous pilot study.

The present study is designed as a randomised-controlled study investigating the effect of post-coercion review.

DETAILED DESCRIPTION:
The present study aims at exploring the impact of a standardized post-coercion review session of coercive measures that took place in the psychiatric inpatient setting in reducing the use of coercive measures and the subjective perception of coercion. It is well known that coercive measures have a major negative impact on the health, well-being and the course of treatment of patients suffering from mental health issues. Many interventions have been implemented in the last years to reduce the use of coercion and limit its consequences.

The investigators developed a standardized post-coercion review intervention. This session takes place as soon as possible after the concerned coercive measure and is moderated by a member of staff who has not been involved in the use of coercion. Other persons involved are the patient, a staff member who took the decision leading to the use of the coercive measure, and a one of the patient's relatives. The guidelines define important themes and questions that should be addressed during the review session. These guidelines have been developed with the help of psychiatrists, nurses and a peer worker.

Hypothesis is that the use of this standardized intervention can reduce the use of subsequent coercive measures and level of perceived coercion, prevent the development of post-traumatic symptoms, help preserving a trustful therapeutic relationship and positively change the attitude of staff regarding the use of coercion. This intervention has been proven to be well accepted by patients and staff members in a previous pilot study. The methods combine quantitative and qualitative evaluations.

The present study is designed as a randomised-controlled study investigating the effect of post-coercion review.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient
* Subject to coercive measure (seclusion, restraint, forced medication)
* Diagnosis of a psychotic disorder (ICD-10: F1x.5, F2x, F31.x).
* Written and informed consent.

Exclusion Criteria:

* Inability to provide informed consent
* Hospital stay < 24h

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Objective coercive measures | At the time of discharge from the hospital by every included patient, up to 6 months
  Number of coercive measures (seclusion, restraint, forced medication)

SECONDARY OUTCOMES:
Subjective experience of coercion (1) | At the time of discharge from the hospital by every included patient, up to 6 months
  Subjective experience coercion assessed by the German version of the Perceived Coercion Subscale (PCS) of the MacArthur Admission Experience Survey (AES). The AES comprises 16 dichotomous items (yes-no answers) divided in 4 subscales. The PCS comprises 5 items. A higher score (range 0-5) indicates a high level of perceived coercion.
Subjective experience of coercion (2) | At the time of discharge from the hospital by every included patient, up to 6 months
  Subjective experience coercion assessed by the Coercion Ladder (CL). The CL is an analog scale ranging from 1 to 10 and assessing the level pf perceived coercion. Higher values indicate a higher level of perceived coercion.
Subjective experience of coercion (3) | At the time of discharge from the hospital by every included patient, up to 6 months
  Subjective experience coercion assessed by the German version of the Coercion Experience Scale (CES). The CES is a scale used to measure the impact of coercive measures. It comprises 29 items related to perceived stressors during a coercive intervention with a 5-point Likert-scale. A total score is used with higher values indicating higher perceived coercion.
Quality of the therapeutic relationship | At the time of discharge from the hospital by every included patient, up to 6 months
  Evaluation of the quality of the therapeutic relationship assessed by the German version of the Work Alliance Inventory-Short Form (WAI-SR). The WAI comprises 12 items divided into 3 subclass (goal, task, bond). each subscale comprises 4 items with a 5-point Likert-scale. The score range for each subscale ranges from 5 to 20. Higher scores indicate a better therapeutic alliance.
Post-traumatic symptoms (1) | At the time of discharge from the hospital by every included patient, up to 6 months
  Development of post-traumatic symptoms assessed by the German version of the Peri-Traumatic Distress Inventory (PDI). The PDI assesses the reactions during the traumatic event. It comprises 13 items with a 0-4 Likert-scale. Scores of all items are summed up and so the total score ranges from 0 to 52. A score higher than 26 indicates a high risk of developing a post traumatic stress disorder.
Post-traumatic symptoms (2) | At the time of discharge from the hospital by every included patient, up to 6 months
  Development of post-traumatic symptoms assessed by the German version of the Impact of Events Scale Revised (IES-R). The IES-R comprises 22 items with a Likert-scale ranging from 0 to 5. Items are divided into 3 sub scales (Intrusion (7 items), Avoidance (8 items), and Hyperarousal (7 items)). Scores for each sub scales are built by adding the answers to each item. Higher scores indicate a higher level of symptoms. The probability of post traumatic stress disorder (PTSD) is assessed using a formula developed by the German translators: X = (-0,02 x intrusion) + (0,07 x avoidance) + (0,15 x hyperarousal) - 4,36. Scores >0 indicate the probable presence of PTSD.

CONTACTS AND LOCATIONS:
Overall Officials: PD Dr. med. Montag, Study Chair — Charité; Dr. med. Mahler, Study Chair — Charité; Dr. med. Wullschleger, Principal Investigator — Charité
Locations (6):
- Germany (6):
  - Psychiatrische Universitätsklink der Charité - SHK, Mitte, State of Berlin
  - Vivantes Klinikum am Urban, Berlin
  - Vivantes Wenckebach-Klinikum, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - Alexianer Krankenhaus Hedwigshöhe, Berlin
  - St. Joseph Krankenhaus Weißensee, Berlin

REFERENCES:
- [Derived] Wullschleger A, Vandamme A, Mielau J, Renner L, Bermpohl F, Heinz A, Montag C, Mahler L. Effect of standardized post-coercion review session on symptoms of PTSD: results from a randomized controlled trial. Eur Arch Psychiatry Clin Neurosci. 2021 Sep;271(6):1077-1087. doi: 10.1007/s00406-020-01215-x. Epub 2020 Nov 24. PMID 33231771